CLINICAL TRIAL: NCT01442155
Title: An Open Label Study of the Effect of Adjuvant Treatment With Capecitabine in Combination With Oxaliplatin on Disease-Free Survival in Patients With Stage III Colon Cancer
Brief Title: An Observational Study of Adjuvant Treatment With Capecitabine (Xeloda) in Combination With Oxaliplatin in Participants With Stage III Colon Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25526
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Results first posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-05

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Adjuvant setting; Capecitabine; Oxaliplatin
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Capecitabine + Oxaliplatin: Participants with stage lll colon cancer, who were starting adjuvant chemotherapy with capecitabine in combination with oxaliplatin according to standard of care.
  Interventions: Drug: Capecitabine; Biological: Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine — Administered according to the Summary of Product Characteristics.
  Other Names: Xeloda
Biological: Oxaliplatin — Administered according to the Summary of Product Characteristics.

SUMMARY:
This observational study evaluates the efficacy and safety of capecitabine in combination with oxaliplatin in the adjuvant setting in participants with Stage III colon cancer. Data were collected from each participant for up to 36 months or until disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Treatment in line with the currently approved indication in the Summary of Product Characteristics

Exclusion Criteria:

* Contraindications according to the current Summary of Product Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Stage III colon cancer
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2011-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Slovakia (8):
  - Banská Bystrica
  - Bratislava
  - Košice
  - Martin
  - Nitra
  - Poprad
  - Prešov
  - Ružomberok

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were screening failures. 74 participants were assigned to the study and treated with study drug.
Period: Overall Study
Arm/Group | Capecitabine + Oxaliplatin
Started | 74
Completed | 9
Not Completed | 65
Not completed — Complete remission | 35
Not completed — Recurrence | 26
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine + Oxaliplatin
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Disease-Free Survival (Time to Event)
Description: Disease free survival was measured as the time from the date of randomization until the date of first event (recurrence of colon cancer, or death due to any cause).
Time Frame: Up to 3 years
Population: Intent-to-treat (ITT) population included all participants treated with at least one dose of study drug. Here, number of participants analyzed is number evaluable for efficacy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine + Oxaliplatin
Number analyzed (Participants) | 67
months | 25 [15.1 to 34.9]

2. Secondary Outcome: Safety: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to 3 years
Population: Safety population included all participants treated with at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine + Oxaliplatin
Number analyzed (Participants) | 74
percentage of participants | 39.19

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Capecitabine + Oxaliplatin
Serious Adverse Events (participants affected / at risk) | 1/74
Other Adverse Events (participants affected / at risk) | 23/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine + Oxaliplatin (N=74)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine + Oxaliplatin (N=74)
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Diarrhea (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 5
Neuropathy peripheral (Nervous system disorders) | 7
Paresthesia (Nervous system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.